CLINICAL TRIAL: NCT02230384
Title: The Development of of A Novel Therapeutic to Aid Tobacco Smoking Cessation in Persons With Schizophrenia or Schizoaffective Disorder
Brief Title: Novel Smoking Cessation Drug for Schizophrenia
Acronym: TRENDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: K.N. Roy Chengappa (Other)
Collaborators: University of Pittsburgh (Other); National Institutes of Health (NIH) (NIH); Virginia Commonwealth University (Other)
Responsible Party: Sponsor-Investigator, K.N. Roy Chengappa, Professor of Psychiatry, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PRO14060338; UH3TR000958 (NIH)
Record Dates: First submitted 2014-07-24; First posted 2014-09-03 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Smoking Cessation
Keywords: Attempt at Smoking Cessation; Schizophrenia or Schizoaffective disorder; Novel nicotinergic drug
MeSH Terms: conditions — Smoking Cessation; Schizophrenia; Psychotic Disorders | interventions — JNJ-39393406

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active JNJ Drug (Experimental): 200 mg (100 mg b.i.d.) Active JNJ Drug used to assess quitting for one week, as part of crossover design. This JNJ experimental compound has NO name, just a company number.
  Interventions: Drug: Active JNJ Drug; Drug: Placebo Pill
- Placebo Pill (Experimental): Placebo pill used for one week quit attempt, as part of crossover design.
  Interventions: Drug: Active JNJ Drug; Drug: Placebo Pill

INTERVENTIONS:
Drug: Active JNJ Drug — 200 mg/day (100 mg b.i.d.) of Active JNJ Drug will be used for one week while attempting to briefly quit smoking on Mon-Fri of that week
  Other Names: JNJ-39393406
Drug: Placebo Pill — Placebo pill will be taken daily to assess ability to briefly quit smoking on Mon-Fri for one week

SUMMARY:
The investigators will evaluate effects of a novel drug that improves nicotinergic receptor function vs. placebo on short-term smoking abstinence in smokers with schizophrenia who have a high interest in quitting. The investigators predict that the novel drug will increase days of abstinence, compared with placebo, identifying potential evidence of efficacy for smoking cessation in smokers with schizophrenia.

The investigators will also assess if this new drug decreases nicotine withdrawal, craving, and cognitive impairment during early abstinence, as well as evaluate adverse effects.

DETAILED DESCRIPTION:
Objective:

This is a Proof of Concept study planned over nearly 2 years to determine the potential efficacy of a novel drug for smokers with schizophrenia.

This study will assess 60 smokers with a diagnosis of either schizophrenia or schizoaffective disorder with high quit interest on their ability to quit during a week-long attempt to abstain while receiving a novel drug vs. placebo, using a within-subjects cross-over design.

Research Plan:

Active drug or placebo will be provided to participants in double-blind fashion.

Study participation will last 6 weeks after subjects enter the study following the screening and physical exam sessions (about 8 weeks total). Participants will engage in two identical study phases, each involving visits over 3 weeks and varying only in whether active drug or placebo is administered. The 3 weeks will involve: baseline visits, dose run-up (week 2), and week 3 (for abstinence assessments). The first week of each period will be a baseline week in which they smoke normally without any medication. During week 2, subjects will begin the dose run-up of active drug or placebo, increasing over 4 days from 1 tablet of 50 mg once daily to 100 mg b.i.d. (two 50 mg tablets twice/day), which will continue through the second and third weeks. Active drug or placebo will be administered in counter-balanced order in a cross-over design. During week 3, subjects will be instructed to try to abstain on each day, i.e. Mon-Friday. Most visits will last 60 mins and involve psychiatric assessments (including psychopathology and neurological and other side effects) ratings, providing an expired breath carbon monoxide (CO) measure that assesses smoking exposure in the past 24 hrs, as well as completing brief self-report measures of craving, withdrawal, and mood. On week 3 of each phase, one visit will involve cognitive testing. On Fri of week 3, subjects will discontinue all medication and resume ad lib smoking prior to the next study period, involving the same 3-week procedure (but with the other medication condition): baseline, dose run-up, full dose administration plus abstinence assessment. Note that active medication will be taken during only one period, with placebo taken during the other period. Pill counts will be used to measure adherence.

Primary and secondary dependent measures are described separately in this report.

Psychopathology will be assessed using standard rating scales to evaluate psychoses and general psychopathology and severity of illness ratings, and suicide rating scales. These and clinical impressions of patients in the study will assist in monitoring for stability or worsening of psychoses or suicidal behavior and/or the need to exit patients from the study.

Laboratory and EKG monitoring at the beginning and end of the study will also be part of the subject safety procedures.

Patients will be offered their choice of one of the FDA approved smoking cessation agents, i.e. nicotine replacement therapy, bupropion or varenicline for a 3-month period upon completion of the study. If patients decline open-label smoking cessation participation, they will be requested to come in for one post-study visit, 14 ± 4 days later. At the first post-study visit, if there are no adverse events, their participation will end.

Methods:

The novel drug or placebo will be administered double-blind in counter-balanced order in a cross-over design. This is not a clinical trial that assesses long term smoking cessation but a within-subjects comparison of the short-term effects of this drug on abstinence and abstinence symptoms over a week-long period, relative to placebo.

Significance:

This study addresses an important question of whether the novel drug shows potential efficacy for smoking cessation, relative to placebo, in smokers with schizophrenia. This procedure could have enormous implications for accelerating the development of this medication and similar compounds to help people quit smoking by increasing the efficiency of early medication evaluation.

ELIGIBILITY:
Inclusion Criteria: List the specific criteria for inclusion of potential subjects.

* Men or women of any race, ages 18 to 65 years, (≥18 years, ≤ 66 years)
* Willing to provide written informed consent
* MINI (Sheehan et al 1998, 2008) chart and/or clinician consensus affirmed DSM IV TR or (DSM -V) diagnoses of schizophrenia or schizoaffective disorder.
* Patients whose PANSS total scores have been stable for ≥ 4 weeks (clinician and/or subject affirmed) and at ≤ 70
* No recent ( ≤ 3months) hospitalization, aggression, or suicidal attempts
* Stable doses of antipsychotic medication, ≥ 4 weeks

Smoking Inclusion Criteria:

* Smoke ≥ 5 cigarettes/day
* Smoking cigarettes ≥ 1 year

Exclusion Criteria:

Smoking/Nicotine Exclusions:

* Use of smokeless tobacco or snuff or chewing tobacco
* Use of e-cigarettes, or any non-tobacco nicotine products (e.g. nicotine gum, lozenges, patch, etc.)
* Current enrollment or plans to enroll in another smoking cessation program. (Bupropion use for depression will be assessed on a case by case basis)

Alcohol/Illicit Substance Exclusion Criteria:

* Recent alcohol or substance dependence (≤ 3 months)
* Current alcohol consumption that exceeds 15 standard drinks/week or greater than 2 standard drinks daily

Medical Exclusion Criteria:

* Women who are pregnant, planning a pregnancy, or lactating; all female participants shall undergo a pregnancy test at screening and will be excluded if positive.
* Serious or unstable medical disorder within the past 3 months (assessed by the investigators)
* Epilepsy
* Current diagnosis (within last 6-months) of abnormal cardiac rhythms; unstable cardiovascular disease e.g. stroke, myocardial infarction in the last 6 months
* Evidence impaired liver function test (LFT) defined as serum glutamate oxaloacetate transaminase (SGOT) (AST) or serum glutamate pyruvate transaminase (SGPT) (ALT) or alkaline phosphatase greater than 1x the upper limit of normal, or bilirubin 1x the upper limit of normal
* Evidence of kidney failure defined as: Serum creatinine > 1.8 mg/dl for males and 1.6 mg/dl for females.
* Any subject with a history of hematological cancers examples: leukemia, lymphoma etc. will be excluded.
* Any clinically significant hematological laboratory abnormality (chronic low-grade laboratory values just above or below the reference range that are without clinical significance will be permitted) will be grounds for exclusion.

Medication Exclusion Criteria:

* Current use or recent discontinuation (within last 14-days) of the following medications: any form of smoking cessation medication (Bupropion except when used for Depressive Disorders on a case by case basis, Varenicline, NRT); and (b) opiate-containing medications for chronic pain. Potent CYP 3A4 inhibitors will be reviewed for exclusion, see below.
* In view of novel drug being a moderate CYP3A4 inhibitor, any subjects receiving the following narrow therapeutic index CYP3A4 substrates will be excluded: Alfentanil, astemizole, cisapride, cyclosporine, dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, sirolimus, tacrolimus, terfenadine.
* In view of the impact of clozapine on smoking cessation, patients receiving clozapine will be excluded.
* Stable medical conditions examples: hypertension, diabetes, dyslipidemia etc that are treated and ongoing and patients are not receiving the exclusionary drugs noted above will be considered for inclusion on a case by case basis.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-12-16 (Actual); Study Completion 2017-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K.N. Roy Chengappa, MD, Principal Investigator — Western Psychiatric Institute and Clinic - UPMC
Locations (1):
- Western Psychiatric Institute and Clinic and affilated sites, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Active JNJ Drug Then Placebo: 200 mg (100 mg b.i.d.) Active JNJ Drug used to assess quitting for one week, as part of crossover design. This JNJ experimental compound has NO name, just a company number.
  Active JNJ Drug: 200 mg/day (100 mg b.i.d.) of Active JNJ Drug will be used for one week while attempting to briefly quit smoking on Mon-Fri of that week
  Placebo Pill: Placebo pill will be taken daily to assess ability to briefly quit smoking on Mon-Fri for one week
- Placebo Pill Then Active JNJ Drug: Placebo pill used for one week quit attempt, as part of crossover design.
  Active JNJ Drug: 200 mg/day (100 mg b.i.d.) of Active JNJ Drug will be used for one week while attempting to briefly quit smoking on Mon-Fri of that week
  Placebo Pill: Placebo pill will be taken daily to assess ability to briefly quit smoking on Mon-Fri for one week
Period: Phase 1
Arm/Group | Active JNJ Drug Then Placebo | Placebo Pill Then Active JNJ Drug
Started | 30 | 32
Completed | 29 | 31
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1
Period: Phase 1 Wash Out
Arm/Group | Active JNJ Drug Then Placebo | Placebo Pill Then Active JNJ Drug
Started | 29 | 31
Completed | 29 | 31
Not Completed | 0 | 0
Period: Phase 2 - Switch
Arm/Group | Active JNJ Drug Then Placebo | Placebo Pill Then Active JNJ Drug
Started | 29 | 31
Completed | 26 | 30
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 2 | 0
Period: Phase 2 Wash Out
Arm/Group | Active JNJ Drug Then Placebo | Placebo Pill Then Active JNJ Drug
Started | 26 | 30
Completed | 26 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active JNJ Drug Then Placebo | Placebo Pill Then Active JNJ Drug | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 32 | 62
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.06 (11.31) | 46.31 (10.97) | 46.19 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 18 | 19 | 37
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 32 | 62

OUTCOME MEASURES:

1. Primary Outcome: Quit Status
Description: Complete abstinence from smoking for 24 hr, assessed daily from Mon-Fri for just one week. This same Mon-Fri procedure for one week (only) is done for both drug phases (Number of days abstinent per each quit week)
  Numbers reported are collapsed across medication conditions for each medication order.
Time Frame: Daily - Mon-Fri during the quit week in each phase
Population: All participants who completed Phase 1 and Phase 2 of the of the study were included in the analysis.
Measure: Mean (Standard Error); unit: days abstinent
Groups:
- Active JNJ Drug: Period during which participants received Active JNJ Drug: 200 mg/day (100 mg b.i.d.)
- Placebo Pill: Period during which Participants received Placebo pill: 200 mg/day (100 mg b.i.d.)
Arm/Group | Active JNJ Drug | Placebo Pill
Number analyzed (Participants) | 56 | 56
days abstinent | 0.46 (0.151) | 0.54 (0.173)

2. Secondary Outcome: Withdrawal When Quit
Description: Severity of withdrawal symptoms will be assessed with standard self-report measures each day during the quit week only of each phase. Data will be analysed when quit criteria were met. Scale used was the Minnesota Nicotine Withdrawal Scale (MNWS), ranging from 0 to 100, with higher scores indicating greater levels of withdrawal symptoms. The MNWS was completed 5 times for each participant during the quit week of each phase. The mean score was used to aggregate across visits.
Time Frame: during each quit week
Population: Participants who met CO < 5 ppm quit criterion.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- JNJ Drug: 200 mg (100 mg b.i.d.) Active JNJ Drug used to assess quitting for one week, as part of crossover design. This JNJ experimental compound has NO name, just a company number.
  Active JNJ Drug: 200 mg/day (100 mg b.i.d.) of Active JNJ Drug will be used for one week while attempting to briefly quit smoking on Mon-Fri of that week
- Placebo: Placebo pill used for one week quit attempt, as part of crossover design.
  Placebo Pill: Placebo pill will be taken daily to assess ability to briefly quit smoking on Mon-Fri for one week
Arm/Group | JNJ Drug | Placebo
Number analyzed (Participants) | 15 | 15
score on a scale | 11.05 (2.86) | 11.52 (1.77)

3. Secondary Outcome: Cognitive Functions
Description: Performance on standardized cognitive tasks (Continuous Performance Task) to determine potential mechanisms of drug efficacy when CO < 10 smoking reduction criteria was met for both sessions. The Continuous Performance Test provides assesses sustained attention in milliseconds.
Time Frame: Assessed at the end of both treatment phases, i.e., at the end of 3 and 6 weeks.
Population: those who met the CO < 10 smoking reduction criteria at the end of both treatment phases
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | JNJ Drug | Placebo
Number analyzed (Participants) | 6 | 6
milliseconds | 519 (37) | 505 (29)

4. Secondary Outcome: Monitoring of Psychiatric Symptoms Including Psychopathology
Description: Psychiatric symptoms using Positive and Negative Syndrome Scale (PANSS) will be conducted at each visit in each 3 week phase of the study
  PANSS - Positive and Negative Syndrome Scale. Min value 30, Max value 210, higher scores are worse outcome.
  The mean score was used to aggregate across visits.
Time Frame: Once at every scheduled visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active JNJ Drug | Placebo Pill
Number analyzed (Participants) | 56 | 56
score on a scale | 42.23 (7.79) | 42.26 (7.63)

5. Secondary Outcome: Number of Participants That Met Criteria for Treatment Emergent Suicidal Ideation or Behavior
Description: CSSRS: Columbia Suicide Severity rating Scale. The scale assesses treatment emergent suicidal ideation and/or behavior categorically as a YES/NO response (no min/max score). "No" responses indicate ideation/behaviors did not emerge "Yes" responses indicate there were ideation or behaviors We are reporting the number of participants that met criteria for suicidal ideation or behavior, based on their CSSRS assessment
Time Frame: Every visit up to six weeks. It is only significant when there is a positive response "Yes"
Measure: Count of Participants; unit: Participants
Groups:
- JNJ Drug: 200 mg (100 mg b.i.d.) Active JNJ Drug used to assess quitting for one week, as part of crossover design. This JNJ experimental compound has NO name, just a company number.
  Active JNJ Drug: 200 mg/day (100 mg b.i.d.) of Active JNJ Drug will be used for one week while attempting to briefly quit smoking on Mon-Fri of that week
  Placebo Pill: Placebo pill will be taken daily to assess ability to briefly quit smoking on Mon-Fri for one week
- Placebo: Placebo pill used for one week quit attempt, as part of crossover design.
  Active JNJ Drug: 200 mg/day (100 mg b.i.d.) of Active JNJ Drug will be used for one week while attempting to briefly quit smoking on Mon-Fri of that week
  Placebo Pill: Placebo pill will be taken daily to assess ability to briefly quit smoking on Mon-Fri for one week
Arm/Group | JNJ Drug | Placebo
Number analyzed (Participants) | 56 | 56
Participants | 0 | 0

6. Secondary Outcome: Number of Participants That Had Treatment Emergent Clinically Significant Abnormal Lab Results
Description: Routine safety labs (included liver and renal labs) were done at baseline, Visit 9, and Visit 18 to determine whether there were treatment emergent clinically significant changes in any of the laboratory parameters. (no subject with abnormal labs at baseline were enrolled in the study) In addition, liver and renal labs were drawn at Visit 4 and Visit 13 to assess for treatment emergent, clinically significant abnormal liver and renal functions.
  The reported results in the data table below show the number of subjects that had treatment emergent clinically significant abnormal lab results at any of the time points.
  If labs were not within the normal range, they were reviewed by the physician investigators to determine whether they were clinically significant.
Time Frame: Weeks 0, 2, 3, 5, 6
Population: Intent to treat population (all participants who received at least one dose of intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Active JNJ Drug Then Placebo | Placebo Pill Then Active JNJ Drug
Number analyzed (Participants) | 26 | 30
Participants
  Liver and Renal Labs Only Wk 2 | 0 | 0
  Routine Labs (including Liver and Renal) Week 3 | 0 | 0
  Liver and Renal Labs Only Wk 5 | 0 | 0
  Routine Labs (including Liver and Renal) Week 6 | 0 | 0

7. Secondary Outcome: The Number of Participants Who Had Treatment Emergent Clinically Significant EKG Results
Description: EKG measures were done at the screening visit and at the end of study to determine whether there were treatment emergent clinically significant changes in the EKG parameters.
  No subjects with abnormal EKGs at baseline were enrolled in the study The data table below shows the number of subjects with clinically significant abnormal EKG results at the end of the study.
Time Frame: Baseline (Week 0) and end of study (week 6)
Population: Intent to treat population (all participants who received at least on dose of intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Active JNJ Drug Then Placebo | Placebo Pill Then Active JNJ Drug
Number analyzed (Participants) | 26 | 30
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Cross-Over study, all subjects received both JNJ and Placebo. Tables below reflect whether the event occurred during the receipt of JNJ or during the receipt of placebo.
  62 subjects were randomized, of whom 7 did not complete the study. Of those 7, 3 were exposed to both JNJ and Placebo, 1 was exposed to the JNJ condition only, 2 were exposed to the placebo condition only and 1 was not exposed to either condition. Thus 60 subjects were exposed to JNJ and 61 subjects were exposed to placebo.
Groups:
- JNJ Drug: Period during which participants received Active JNJ Drug: 200 mg/day (100 mg b.i.d.)
- Placebo: Period during which Participants received Placebo pill: 200 mg/day (100 mg b.i.d.)
Arm/Group | JNJ Drug | Placebo
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/61
Serious Adverse Events (participants affected / at risk) | 1/60 | 2/61
Other Adverse Events (participants affected / at risk) | 30/60 | 36/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JNJ Drug (N=60) | Placebo (N=61)
aspiration/pneumonia (Immune system disorders) | 0 (0) | 1 (1)
acute diastolic congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1)
persistent vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — This event occurred during the wash out period following having the active JNJ drug
vaginal bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) — This event occurred during the wash out period following having the active JNJ drug
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JNJ Drug (N=60) | Placebo (N=61)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 8 (10)
Nausea (Gastrointestinal disorders) | 4 (5) | 7 (8)
Headache (Nervous system disorders) | 3 (3) | 5 (7)
Somnolence (Nervous system disorders) | 5 (5) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (5) | 2 (3)
Muscle pain/soreness (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Cold/nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Fever (General disorders) | 4 (4) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes